CLINICAL TRIAL: NCT00568698
Title: A Pilot Therapeutic Trial Using Hydroxyurea in Type I Spinal Muscular Atrophy Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SU-11012007-783; 78811; NCT00083746 (obsolete NCT alias)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Hydroxyurea

ARMS (2):
- Hydroxyurea (Experimental)
  Interventions: Drug: Hydroxyurea
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo to match hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea
  Arms: Hydroxyurea
Drug: Placebo to match hydroxyurea
  Arms: Placebo

SUMMARY:
The objectives of this trial are: to establish a safety profile for use of Hydroxyurea in children with Type I Spinal Muscular Atrophy; to identify reliable outcome measures for HU treatment in Type I SMA; and to detect the clinical efficacy of HU treatment in children with Type I SMA.

DETAILED DESCRIPTION:
SMA is a neuromuscular disorder characterized by degeneration of spinal cord motor neurons and muscular atrophy. SMA is classified into three clinical subtypes according to the severity and age of onset (Types I, II and III). Type I SMA (also called severe, infantile or acute SMA, or Werdnig-Hoffman disease) is the most severe phenotype. The onset of symptoms is within the first 6 months of life, and weakness of intercostal muscles and lack of airway protection lead to respiratory insufficiency and aspiration pneumonia, often resulting in early infant death.

In our laboratory, our preliminary results indicate that HU treatment significantly increases both SMN mRNA expression and intact SMN protein levels in vitro. These data confirm previous observations that in vitro treatments of SMA lymphocytes with hydroxyurea resulted in augmentation of the SMN2 gene expression in a dose and time related manner. Based on these exciting pre-clinical data, coupled with the well-documented side-effect profile of HU in children, we are conducting a pilot clinical trial using HU in children with Type I SMA. This clinical trial study is intended to establish the safety profile in children with Type I SMA; to identify reliable outcome measures; and to detect the possible clinical efficacy of HU treatment in children with Type I SMA.

ELIGIBILITY:
Inclusion Criteria:1. Laboratory confirmation of a homozygous deletion or mutation of the SMN1 gene 2. Clinical Diagnosis of Type I SMA (never achieved independent sitting) 3. Onset of disease before the age of 6 months 4. Enrollment in study within 6 months of diagnosis Exclusion Criteria:1. Known hematological disorders, such as chronic anemia (defined as platelet count less than 100,000/mm^3) in two contiguous measures in two weeks 2. Severe systemic disorders such as congenital heart disease, other major birth defects involving internal organs, or severe birth asphyxia 3. Participation in SMA clinical trials for other experimental drugs 4. Requiring continuous respiratory support before the initiation of HU treatment

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2004-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ching H. Wang, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data are presented for all participants because data relating to arm assignment are no longer accessible; the Principal Investigator (PI) has left institution and all efforts to locate the data have been exhausted.
Groups:
- All Participants: Participants received hydroxyurea, or placebo to match hydroxyurea.
Period: Overall Study
Arm/Group | All Participants
Started | 29
Completed | 18
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: Data are presented for all participants because data relating to arm assignment are no longer accessible; the PI has left institution and all efforts to locate the data have been exhausted.
Arm/Group | All Participants
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Safety: Frequency of Adverse Events/Lab Abnormalities
Time Frame: Up to 8 years, 1 month
Population: Data for this outcome measure are no longer accessible; the PI has left institution and all efforts to locate the data have been exhausted.
Groups:
- Hydroxyurea: Hydroxyurea
- Placebo: Placebo to match hydroxyurea
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Efficacy: Length of Survival (LOS) and Age of Ventilator Dependence (AVD)
Time Frame: Up to 8 years, 1 month
Population: as for outcome 1
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Motor Unit Number Estimation (MUNE)
Time Frame: Up to 8 years, 1 month
Population: as for outcome 1
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Biomarker Assays: SMN Protein and SMN mRNA
Time Frame: Up to 8 years, 1 month
Population: as for outcome 1
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 8 years, 1 month
Description: Adverse events data are no longer accessible; the PI has left institution and all efforts to locate the data have been exhausted.
Arm/Group | Hydroxyurea | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes